CLINICAL TRIAL: NCT00668005
Title: A Randomized, Double-blind, Parallel-group, Plac-controlled Study Evaluating the Efficacy and Safety of Vardenafil Administration for 12 Weeks in a Flexible-dose Regimen Compared to Placebo in Men With Arterial Hypertension and Erectile Dysfunction
Brief Title: Evaluating the Efficacy and Safety of Vardenafil in Subjects With Erectile Dysfunction and Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100539
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Arterial hypertension; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction; Hypertension | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 5mg, 10mg or 20mg taken 1h before sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
Assess efficacy of Vardenafil in patients erectile dysfunction and high blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age, with 6 months or longer diagnosis of ED as defined by NIH Consensus statement,
* Arterial hypertension adequately controlled
* Stable sexual relationship for > 6 month

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2003-02; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Sexual Encounter Profile (SEP), questions 2 and 3 | 12 weeks

SECONDARY OUTCOMES:
International Index of Erectile Function (IIEF) - EF (Erectile Function) domain | 12 weeks
Global Assessment Questionnaire (GAQ) | 12 weeks
Safety and tolerability | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer